CLINICAL TRIAL: NCT04927273
Title: Prevalence of Spine Surgery Navigation Techniques and Availability in Africa: A Cross-sectional Study
Brief Title: Availability of Spine Neuronavigation in Africa
Status: Completed | Type: Observational
Sponsor: Association of Future African Neurosurgeons, Yaounde, Cameroon (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: AFAN1
Record Dates: First submitted 2021-06-08; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Spine Disease
Keywords: Access; Africa; computer-assisted surgery; neuronavigation; spine surgery
MeSH Terms: conditions — Spinal Diseases | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Surveyed neurological and orthopedic surgeons

SUMMARY:
In this study, the availability of spine neuronavigation in Africa was evaluated. Access to surgical equipment is an important goal of global surgery and global neurosurgery. The study findings show that there are regional differences in access to spine neuronavigation techniques and highlight that the major barriers to increased prevalence are cost and lack of trained personnel.

ELIGIBILITY:
Inclusion Criteria:

* Neurological and orthopedic surgery residents, fellows and consultants working in Africa.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurological and orthopedic surgery residents, fellows and consultants working in Africa.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Availability of neuronavigation | 1 month
  Number of neuronavigation units as discrete unitless counts available at African neurosurgery centers will be collected using an electronic survey

CONTACTS AND LOCATIONS:
Locations (1):
- Association of Future African Neurosurgeons, Yaoundé, Centre Region, Cameroon

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be shared with authorized personnel only.